CLINICAL TRIAL: NCT02604082
Title: Comparison of Three Technical Airway Clearance in Mechanical Ventilated Patients
Acronym: ClearanceMV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 11-0367
Record Dates: First submitted 2015-11-06; First posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Mucociliary Clearance Defect; Physical Disability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vibocompression (VB) (Active Comparator): Grup 1 - Vibrocompression: Is a physical therapy technique, that aims to clear the airways of patients on mechanical ventilation. Through the thoracic compression during expiration
  Interventions: Other: Vibrocompression (VB)
- Hyperinflation (HMV) (Active Comparator): Grup 2 - Hyperinflation with Mechanical ventilator: Is a physical therapy technique, that aims to clear the airways of patients on mechanical ventilation. Through the increase in inspiratory pressure ventilator .
  Interventions: Other: Hyperinflation (HMV)
- HMV+VB (Experimental): Grup 3 - Hyperinflation with mechanical ventilator and vibrocompression:Is a physical therapy technique, that aims to clear the airways of patients on mechanical ventilation. Through the thoracic compression during expiration and the increase in inspiratory pressure ventilator.
  Interventions: Other: HMV+VB

INTERVENTIONS:
Other: Vibrocompression (VB) — Vibrocompression is a physical therapy technique, that aims to clear the airways of patients on mechanical ventilation (MV)
  Other Names: Techinique of physical therapy
  Arms: Vibocompression (VB)
Other: Hyperinflation (HMV) — Hyperinflation technique with mechanical ventilator which aims to clear the airways of patients on mechanical ventilation
  Other Names: Techinique of physical therapy
  Arms: Hyperinflation (HMV)
Other: HMV+VB — Association between Vibrocompression and Hyperinflation with mechanical ventilator
  Other Names: Techinique of physical therapy
  Arms: HMV+VB

SUMMARY:
Randomized clinical trial, conducted in the Intensive Care Unit of the Hospital de Clinicas de Porto Alegre from october 2011 until november 2015 .

DETAILED DESCRIPTION:
Objective: To compare the effectiveness of techniques: vibrocompression (G1), hyperinflation with mechanical ventilation (G2) vibrocompression + hyperinflation with mechanical ventilation (G3) in the amount of aspirated secretions, mechanical ventilator time, incidence of ventilator-associated pneumonia , reintubation tracheal and mortality in mechanical ventilator. Primary outcome: weight in grams of the aspirated secretions. Secondary outcome: hemodynamic and pulmonary parameters: heart rate, respiratory rate, mean arterial pressure, peripheral arterial oxygen saturation; peak inspiratory pressure, tidal volume; dynamic compliance ; mechanical ventilator time; reintubation tracheal; Incidence of ventilator-associated pneumonia and mortality in mechanical ventilator.

ELIGIBILITY:
Inclusion Criteria:

* In mechanical ventilation for a period of 24-72 h
* End-expiratory pressure (PEEP) lower 10 cm of water.
* Lower noradrenaline doses of 0.5mg / kg / minute for an average greater than or equal blood outstrips 60 mmHg.

Exclusion Criteria:

* Pneumothorax and hemothorax undrained
* Subcutaneous emphysema
* Osteoporosis
* Acute respiratory distress syndrome - (ARDS)
* Fractures of ribs
* Obese ( BMI greater than 35)
* Mechanical ventilator with higher peak pressures 40 cm of water.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-09; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Weight in grams of the pulmonary secretions | up to 24 weeks.

SECONDARY OUTCOMES:
Time mechanical ventilator (MV) in days | Through study completion, an average of 3 years.
Reintubation tracheal in percentage in the last 24 hours | Through study completion, an average of 3 years.
Incidence of ventilator-associated pneumonia in percentage | Through study completion, an average of 3 years.
Mortality in the MV in percentage | Through study completion, an average of 3 years.
Heart Rate | up to 24 weeks.
Respiratory frequency | up to 24 weeks
Peripheral oxygen saturation in percentage | up to 24 weeks
Tidal volume in milliliters | up to 24 weeks
Peak inspiratory pressure in centimeters of water | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Silvia R Rios Vieira, Dr, Principal Investigator — HCPorto Alegre, Rio Grande do Sul - Brazil

REFERENCES:
- [Result] Naue Wda S, Forgiarini Junior LA, Dias AS, Vieira SR. Chest compression with a higher level of pressure support ventilation: effects on secretion removal, hemodynamics, and respiratory mechanics in patients on mechanical ventilation. J Bras Pneumol. 2014 Jan-Feb;40(1):55-60. doi: 10.1590/S1806-37132014000100008. PMID 24626270